CLINICAL TRIAL: NCT00321178
Title: Randomised Trial for Early Lesions Caused by M. Ulcerans - Comparison Between 8 Weeks Streptomycin and Rifampicin (SR), or 4 Weeks SR Followed by 4 Weeks R Plus Clarithromycin
Brief Title: BURULICO Drug Trial Study Protocol: RCT SR8/SR4+CR4, GHANA
Acronym: BURULICO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Prof TS van der Werf, UMCG, University of Groningen, the Netherlands
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BURULICODRUGTRIAL; EU FP6 2003-INCO-Dev2-015476
Record Dates: First submitted 2006-05-02; First posted 2006-05-03 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-04

CONDITIONS: Buruli Ulcer; Mycobacterium Ulcerans
Keywords: Mycobacterium ulcerans; Buruli ulcer; Ghana; randomized comparison; streptomycin; rifampicin; clarithromycin
MeSH Terms: conditions — Buruli Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SR4/CR4 (Experimental): after 4 weeks of standard treatment with streptomycin and rifampicin, patients in the experimental arm switch to oral treatment consisting of rifampicin and clarithromycin
  Interventions: Drug: SR4 - switch to CR4
- SR8 (Active Comparator): standard treatment consisting of 8 weeks of streptomycin and rifampicin
  Interventions: Drug: SR4 - switch to CR4

INTERVENTIONS:
Drug: SR4 - switch to CR4 — switch to oral treatment after 4 weeks SR 'standard' therapy
  Other Names: clarithromycin: Clacid

SUMMARY:
The standard for treatment Buruli ulcer disease (BUD) used to be surgery but the WHO now advises streptomycin (S, 15 mg/kg daily, intramuscularly) and rifampicin (R,10 mg/kg daily) along with surgery. This preliminary advice was based on observations in 21 patients with pre-ulcerative lesions of BUD, who were given daily SR treatment for varying periods of time. In patients treated with SR for at least 4 weeks, M. ulcerans could no longer be cultured from excised lesions. SR has been introduced without a formal evaluation or comparison with other treatments have been conducted or published, but the impression is that this treatment is beneficial and may cure BUD without additional surgical management.

This study protocol evaluated the hypothesis that early, limited lesions of BUD(pre-ulcerative or ulcerated lesions, ≤ 10 cm maximum diameter), can be healed without recurrence using antimycobacterial drug therapy, without the need for debridement surgery.

In endemic regions in Ghana, patients will be actively recruited and followed if ≥ 5 years of age, and with early (i.e., onset < 6 months) BUD.

* consent by patients and / or care givers / legal representatives
* clinical evaluation, and by
* analysis of three 0.3 cm punch biopsies under local anaesthesia.
* disease confirmation: dry reagent-based polymerase chain reaction (DRB-PCR IS2404)
* randomization: either SR for 8 weeks, or 4 weeks of SR followed by R and clarithromycin (C)
* stratification: ulcerative or pre-ulcerative lesions.

Biopsies processed for histopathology, DRB-PCR-, microscopy, culture, genomic, and sensitivity tests. Lesions assessed regularly for progression or healing during treatment. Drug toxicity monitoring included blood cell counts, liver enzymes and renal tests; and ECG and audiographic tests.

Primary endpoint: healing without recurrence at 12 months follow-up after start of treatment Secondary endpoint: reduction in lesion surface area and/or clinically assessed improvement on completion of treatment, averting the need for debridement surgery.

Recurrences biopsied for confirmation, using PCR, histopathology, and culture. Sample size calculation: 2x74 fully evaluable patients; 80% power to detect a difference of 20 % in recurrence-free cure 12 months after start of treatment between the two groups (60 versus 80%). A Data Safety and Monitoring Board made interim analysis assessments.

DETAILED DESCRIPTION:
Buruli ulcer disease (BUD) is caused by infection with Mycobacterium ulcerans. It usually starts as a small nodule under the skin but may progress to an ulcerative lesion; and eventually large, usually painless ulcers may develop. When it heals - with surgery or without - it may cause severe scarring resulting in disability and deformity. BUD has emerged as an important infectious disease among rural populations in West Africa. The standard treatment used to be surgical excision for all forms and stages. In 2004. The World Health Organisation advised the use of streptomycin (S, 15 mg/kg daily, intramuscularly) and rifampicin (R,10 mg/kg daily) along with surgery. This preliminary advice was based on the observation in 21 patients with pre-ulcerative lesions of BUD, who were given daily SR treatment for varying periods of time. If patients had received such treatment for at least 4 weeks, M. ulcerans could not be cultured again from the lesions that were excised. The treatment has been implemented in areas with poor access to surgical facilities, in Pobe, Benin, and although no formal evaluation or comparison with other treatments have been conducted or published, the impression is that this treatment is probably beneficial and may cure BUD without the need for additional surgical management.

This study protocol was designed to evaluate the hypothesis that early, limited lesions of Buruli ulcer (M. ulcerans disease; pre-ulcerative or ulcerated lesions, less than or equal to 10 maximum diameter), can be healed without recurrence using antimycobacterial drug therapy, without the need for debridement surgery.

In endemic regions in Ghana, active case finding will be followed by accrual of patients

* 5 years of age and over, with
* limited early (i.e., onset less than 6 months) lesions of Buruli ulcer.

After appropriate consent by patients and / or their care givers or legal representatives, patients will be diagnosed both by

* clinical evaluation, and
* by analysis of three punch biopsies (0.3 cm each) under local anaesthesia.

Only patients with confirmation of M. ulcerans disease - presence of dry reagent-based polymerase chain reaction (DRB-PCR) signal with insertion sequence IS2404, were to be randomised to receive either SR for 8 weeks, or 4 weeks of SR followed by oral treatment consisting of R and clarithromycin (C), as allocated by a computer-generated program; patients will be stratified for ulcerative or pre-ulcerative lesions.

Patients who meet the clinical criteria for M ulcerans disease but are PCR negative, will be offered 8 weeks RS treatment, as is presently provisionally recommended by WHO, and will be evaluated separately, according to the protocol for patients allocated to 8 weeks RS treatment. All biopsies from lesions will be subjected to histopathology, DRB-PCR-, microscopy, culture, genomic, sensitivity tests and external quality control in laboratories in Kumasi (KNUST), Hamburg (BNITM), Munich (DITM) and Antwerp (ITM). Lesions will be assessed regularly for progression or healing during treatment. Drug toxicity will likewise be monitored: renal and audiographic tests for S and C, ECG for C, and liver enzymes for R and C, and blood cell counts for C.

The primary endpoint is healing without recurrence at 12 months follow-up after start of treatment Secondary endpoint is reduction in lesion surface area and/or clinically assessed improvement on completion of treatment, averting the need for debridement surgery.

Recurrences will be biopsied for confirmation, using PCR, histopathology, and culture. In all, 200 patients will need to be screened according to protocol, and 2x74 evaluable patients will be randomised based on a power analysis to detect a difference of 20 % in recurrence-free cure 12 months after start of treatment between the two groups (60 versus 80%). A Data Safety and Monitoring Board will make interim analyses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* At least 5 years of age
* A clinical diagnosis of early M. ulcerans disease including:

  * Nodules
  * Plaques and small ulcers with or without oedema and less than or equal to 10cm in maximum diameter
  * Disease duration no longer than six months
  * DRB-PCR positive for M. ulcerans

Exclusion Criteria:

* Treatment with macrolide or quinolone antibiotics, or antituberculous medication, or immunomodulatory drugs including corticosteroids within the previous one month.
* Current treatment with any drugs likely to interact with the study medication, e.g, anticoagulants, cyclosporin, phenytoin, oral contraceptive, and phenobarbitone.
* History of hypersensitivity to rifampicin, streptomycin and or clarithromycin.
* History or having current clinical signs of ascites, jaundice, partial or complete deafness, myasthenia gravis, renal dysfunction (known or suspected), diabetes mellitus, and immune compromise; or evidence for past or present tuberculosis.
* Pregnancy
* Inability to take oral medication or having gastrointestinal disease likely to interfere with drug absorption.
* Excessive alcohol intake.
* Any situation or condition which may compromise ability to comply with the trial procedures.
* Lack of willingness to give informed consent (and/or assent by parent/legal representative).

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2006-05; Primary Completion 2008-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
healing without recurrence and without debridement surgery at 12 months follow-up after start of treatment | 12 months follow-up after start of treatment

SECONDARY OUTCOMES:
reduction in lesion surface area and/or clinically assessed improvement on completion of treatment, averting the need for debridement surgery | during treatment and follow-up x 12 months
adverse events | during treatment and follow-up x 12 months
functional limitations | at end of follow-up (12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Tjip S van der Werf, MD PhD, Principal Investigator — University Medical Centre Groningen, University of Groningen, the Netherlands
Locations (2):
- Ghana (2):
  - Agogo Hospital, Agogo, Ashanti Region
  - Nkawie-Toaso Hospital, Nkawie, Ashanti Region

REFERENCES:
- [Background] van der Werf TS, Stienstra Y, Johnson RC, Phillips R, Adjei O, Fleischer B, Wansbrough-Jones MH, Johnson PD, Portaels F, van der Graaf WT, Asiedu K. Mycobacterium ulcerans disease. Bull World Health Organ. 2005 Oct;83(10):785-91. Epub 2005 Nov 10. PMID 16283056
- [Background] van der Werf TS, van der Graaf WT, Tappero JW, Asiedu K. Mycobacterium ulcerans infection. Lancet. 1999 Sep 18;354(9183):1013-8. doi: 10.1016/S0140-6736(99)01156-3. PMID 10501380
- [Background] Etuaful S, Carbonnelle B, Grosset J, Lucas S, Horsfield C, Phillips R, Evans M, Ofori-Adjei D, Klustse E, Owusu-Boateng J, Amedofu GK, Awuah P, Ampadu E, Amofah G, Asiedu K, Wansbrough-Jones M. Efficacy of the combination rifampin-streptomycin in preventing growth of Mycobacterium ulcerans in early lesions of Buruli ulcer in humans. Antimicrob Agents Chemother. 2005 Aug;49(8):3182-6. doi: 10.1128/AAC.49.8.3182-3186.2005. PMID 16048922
- [Derived] Barogui YT, Klis SA, Johnson RC, Phillips RO, van der Veer E, van Diemen C, van der Werf TS, Stienstra Y. Genetic Susceptibility and Predictors of Paradoxical Reactions in Buruli Ulcer. PLoS Negl Trop Dis. 2016 Apr 20;10(4):e0004594. doi: 10.1371/journal.pntd.0004594. eCollection 2016 Apr. PMID 27097163
- [Derived] Nienhuis WA, Stienstra Y, Abass KM, Tuah W, Thompson WA, Awuah PC, Awuah-Boateng NY, Adjei O, Bretzel G, Schouten JP, van der Werf TS. Paradoxical responses after start of antimicrobial treatment in Mycobacterium ulcerans infection. Clin Infect Dis. 2012 Feb 15;54(4):519-26. doi: 10.1093/cid/cir856. Epub 2011 Dec 7. PMID 22156855
- [Derived] Nienhuis WA, Stienstra Y, Thompson WA, Awuah PC, Abass KM, Tuah W, Awua-Boateng NY, Ampadu EO, Siegmund V, Schouten JP, Adjei O, Bretzel G, van der Werf TS. Antimicrobial treatment for early, limited Mycobacterium ulcerans infection: a randomised controlled trial. Lancet. 2010 Feb 20;375(9715):664-72. doi: 10.1016/S0140-6736(09)61962-0. Epub 2010 Feb 3. PMID 20137805
- See also: Global Buruli ulcer Initiative, World Health organisation — http://www.who.int/buruli/en/
- See also: Kumasi Centre for Collaborative Research, Kwame Nkrumah University of Science and Technology, Kumasi, Ghana — http://www.kccr.de/kccr/
- See also: University Medical Centre Groningen, University of Groningen, the Netherlands — http://www.rug.nl/umcg/index?lang=en